CLINICAL TRIAL: NCT03093233
Title: German-wide Multicenter Analysis of Oral Anticoagulant-associated Intracerebral Hemorrhage - Part Two (RETRACE-II)
Brief Title: Multicenter Analysis of Oral Anticoagulant-associated ICH - Part Two
Acronym: RETRACE-II
Status: Completed | Type: Observational
Sponsor: University of Erlangen-Nürnberg Medical School (Other)
Responsible Party: Sponsor
Other Study IDs: MulticenterAnalysis OAC-ICH-II
Record Dates: First submitted 2017-03-03; First posted 2017-03-28 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2017-03

CONDITIONS: Anticoagulation Associated (VKA & NOAC) Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- VKA- and NOAC-related ICH: 1. Analysis of hematoma enlargement: prevalence, risk factor, associations with therapeutic interventions (in patients with cranial follow-up imaging)
  2. Association of hematoma evacuation surgery with clinical outcomes
  3. Associations of antithrombotic management with ischemic and hemorrhagic complications
  4. Safety of intraventricular fibrinolysis (in patients with severe intraventricular hemorrhage)
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — only descriptive data analysis

SUMMARY:
Intracerebral hemorrhage [ICH] is the most feared complication of oral anticoagulation [OAC], yet therapeutic strategies are limited reflected by overall weak guideline recommendations. Studies investigating acute interventions especially in patients with ICH taking non-vitamin-K-oral-anticoagulants [NOAC] remain inconclusive. Further, acute management issues in OAC-ICH patients (hematoma evacuation surgery, prevention of acute thromboembolic events, intraventricular fibrinolysis) still need to be investigated. Therefore, this observational study (RETRACE-II) represents the follow-up investigation to RETRACE (German-wide Multicenter Analysis of Oral Anticoagulant-associated Intracerebral Hemorrhage, study-period 2006-2010, NCT01829581), now spanning a study-period from 2011 until 2015 with 19 participating tertiary care centers nation-wide in Germany. Data pooling of the two RETRACE studies, altogether including more than 2500 patients treated at 22 centers over a 10 year period will allow statistically appropriate analyses of different outcomes.

DETAILED DESCRIPTION:
Stroke in general is one of the leading causes for death and disability in the industrialized world. Cardiac thrombo-embolisms are the major contributor to ischemic infarction with atrial fibrillation [afib] being the most frequent underlying pathology. As the prevalence of afib is constantly increasing with the ageing population, its established therapy (oral anticoagulation with vitamin-K antagonists [VKA] or non-vitamin-K-oral-anticoagulants [NOAC]) will increase alongside. Therefore, rates of OAC-ICH are expected to increase simultaneously. OAC-ICH is associated with larger ICH-volumes, an increased frequency of hematoma enlargement, and worse clinical outcome as compared to primary spontaneous ICH. Nevertheless, only limited evidence exists regarding acute treatment strategies. For the prevention of hematoma enlargement in VKA-ICH a large observational cohort study (n=1176) for the first time identified a time window (<4h) and INR level (INR<1.3) within which reversal of altered coagulation may show reduced rates of hematoma enlargement (1). For NOAC-ICH only very small sized investigations or case reports are available to address this pressing question - how to reverse anticoagulation in NOAC-ICH. Existing data does not even allow appropriate description of NOAC-ICH patients in terms of hematoma characteristics, re-bleeding rates, neurologic severity or functional outcome. Due to this dilemma and without available antidotes (except for dabigatran) reversal strategies are intensely debated and evidence based guideline recommendations do not exist. Further important treatment approaches in ICH-care such as (i) hematoma evacuation surgery, (ii) early anticoagulation or prophylaxis of systemic thromboembolisms, (iii) intraventricular fibrinolysis, have not been investigated as this growing sub-population (increasing incidence) has been vastly excluded from randomized trials.

Therefore, this observational cohort study (RETRACE-II) will try to strengthen the therapeutic evidence for OAC-ICH treatment by data-assessment of 19 nation-wide tertiary care hospitals in Germany. Patients will be identified from medical records by the diagnosis of ICH and concomitantly present intake of VKA (INR>1.5) or known intake of NOAC during a time period from 20011-2015. Only patients with ICH associated to OAC will be included, other secondary causes i.e. tumors, trauma, vascular malformations or aneurysms etc. will be excluded. Clinical data on demographics, medical history, pre-ICH medication exposures and laboratory results will be obtained by medical charts, institutional databases or prospective registries, supplemented by structured interviews or by review of available medical records at each individual institution. Patient-derived follow-up information will be corroborated by review of pertinent medical records. An estimated total number of greater 1000 patients will be reviewed for this investigation. In detail the following parameters will be evaluated: - prior medical history (including CHADS-VASC-Score, HAS-Bled Score, vascular risk factors), - functional status prior admission (mRS), - neurological admission status (NIHSS, GCS), - imaging characteristics, - time intervals: symptom onset until admission, imaging, therapy initiation, - mode of hemostatic therapy, - acute blood pressure management, - complications (hemorrhagic- or ischemic-events, infectious) and treatment (surgical treatment, mode of antithrombotic treatment or prophylaxis of systemic thromboembolism, intraventricular fibrinolysis, etc.), - mortality rates, - functional outcome (mRS).

Participating Centers (upon Invitation):

Klinikum Bad Hersfeld, Department of Neurology, Germany. HELIOS Klinikum Berlin-Buch, Department of Neurology, Germany. University Hospital Charité Berlin, Department of Neurology, Germany. Klinikum Dortmund, Department of Neurology, Germany. University of Dresden, Department of Neurology, Germany. Asklepios Klinik Hamburg Altona, Department of Neurology, Germany. Heidelberg University Hospital, Department of Neurology, Germany. University of Jena, Department of Neurology, Germany. Klinikum Koblenz, Department of Neurology, Germany. University of Cologne, Department of Neurology, Germany. University of Leipzig, Department of Neurology, Germany. Klinikum der Stadt Ludwigshafen am Rhein, Department of Neurology, Germany. Johannes Wesling Medical Center Minden, Department of Neurology, Germany. University of Münster, Department of Neurology, Germany. Klinikum Nürnberg, , Department of Neurology, Germany. Klinikum Stuttgart, Department of Neurology, Germany. University of Ulm, Department of Neurology, Germany. University of Wuerzburg, Department of Neurology, Germany.

Funding:

This study was partly supported by research grants from the Johannes & Frieda-Marohn Foundation (FWN/Zo-Hutt/2011) and from the ELAN fonds (ELAN 12.01.04.1), University of Erlangen, Germany.

ELIGIBILITY:
Inclusion Criteria:

* VKA-ICH defined as effective use of VKA with an INR-value of >1.5 on hospital admission
* NOAC-ICH defined as known to be on treatment with NOAC at ICH-onset

Exclusion Criteria:

* ICH related to trauma, tumor, arteriovenous malformation, aneurysmal subarachnoid hemorrhage, acute thrombolysis, or other coagulopathies.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Anticoagulation (VKA & NOAC) associated ICH
Sampling Method: Probability Sample
Enrollment: 1369 (Actual)
Dates: Start 2016-01-01 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-08-30 (Actual)

PRIMARY OUTCOMES:
Hematoma enlargement (NOAC- versus VKA-ICH) | 24hour
Intracranial complications (ischemic and hemorrhagic events) | through study period (hospital stay), an average of 14day
Extracranial complications (ischemic and hemorrhagic events) | through study period (hospital stay), an average of 14day
Mortality | at 90 days
Functional outcome (modified Rankin-Scale 4-6) | at 90 days

SECONDARY OUTCOMES:
Systolic blood pressure level in NOAC-ICH | 24hour
Functional outcome (modified Rankin-Scale 4-6) after hematoma evacuation surgery | at 90 days
Functional outcome (modified Rankin-Scale 4-6) according to anticoagulation treatment | at 90 days
Functional outcome (modified Rankin-Scale 4-6) after intraventricular fibrinolysis | at 90 days

CONTACTS AND LOCATIONS:
Overall Officials: Hagen B. Huttner, MD., Principal Investigator — University Hospital Erlangen, Department of Neurology, Germany; Joji B. Kuramatsu, MD., Principal Investigator — University Hospital Erlangen, Department of Neurology, Germany

REFERENCES:
- [Background] Kuramatsu JB, Gerner ST, Schellinger PD, Glahn J, Endres M, Sobesky J, Flechsenhar J, Neugebauer H, Juttler E, Grau A, Palm F, Rother J, Michels P, Hamann GF, Huwel J, Hagemann G, Barber B, Terborg C, Trostdorf F, Bazner H, Roth A, Wohrle J, Keller M, Schwarz M, Reimann G, Volkmann J, Mullges W, Kraft P, Classen J, Hobohm C, Horn M, Milewski A, Reichmann H, Schneider H, Schimmel E, Fink GR, Dohmen C, Stetefeld H, Witte O, Gunther A, Neumann-Haefelin T, Racs AE, Nueckel M, Erbguth F, Kloska SP, Dorfler A, Kohrmann M, Schwab S, Huttner HB. Anticoagulant reversal, blood pressure levels, and anticoagulant resumption in patients with anticoagulation-related intracerebral hemorrhage. JAMA. 2015 Feb 24;313(8):824-36. doi: 10.1001/jama.2015.0846. PMID 25710659
- [Derived] Huttner HB, Gerner ST, Kuramatsu JB, Connolly SJ, Beyer-Westendorf J, Demchuk AM, Middeldorp S, Zotova E, Altevers J, Andersohn F, Christoph MJ, Yue P, Stross L, Schwab S. Hematoma Expansion and Clinical Outcomes in Patients With Factor-Xa Inhibitor-Related Atraumatic Intracerebral Hemorrhage Treated Within the ANNEXA-4 Trial Versus Real-World Usual Care. Stroke. 2022 Feb;53(2):532-543. doi: 10.1161/STROKEAHA.121.034572. Epub 2021 Oct 14. PMID 34645283
- [Derived] Gerner ST, Kuramatsu JB, Sembill JA, Sprugel MI, Hagen M, Knappe RU, Endres M, Haeusler KG, Sobesky J, Schurig J, Zweynert S, Bauer M, Vajkoczy P, Ringleb PA, Purrucker JC, Rizos T, Volkmann J, Mullges W, Kraft P, Schubert AL, Erbguth F, Nueckel M, Schellinger PD, Glahn J, Knappe UJ, Fink GR, Dohmen C, Stetefeld H, Fisse AL, Minnerup J, Hagemann G, Rakers F, Reichmann H, Schneider H, Rahmig J, Ludolph AC, Stosser S, Neugebauer H, Rother J, Michels P, Schwarz M, Reimann G, Bazner H, Schwert H, Classen J, Michalski D, Grau A, Palm F, Urbanek C, Wohrle JC, Alshammari F, Horn M, Bahner D, Witte OW, Gunther A, Hamann GF, Engelhorn T, Lucking H, Dorfler A, Schwab S, Huttner HB. Characteristics in Non-Vitamin K Antagonist Oral Anticoagulant-Related Intracerebral Hemorrhage. Stroke. 2019 Jun;50(6):1392-1402. doi: 10.1161/STROKEAHA.118.023492. Epub 2019 May 16. PMID 31092170